CLINICAL TRIAL: NCT07331090
Title: A Comparative Evaluation of Removable Appliances and Clear Aligners in Terms of Multidimensional Parameters and Their Effects on Phonation in Early Orthodontic Treatments During the Mixed Dentition Period
Brief Title: Evaluation of Removable Appliances and Clear Aligners in Early Orthodontic Treatments During the Mixed Dentition Period
Status: Completed | Type: Observational
Sponsor: Neslihan Atmaca (Other)
Collaborators: Marmara University (Other)
Responsible Party: Sponsor-Investigator, Neslihan Atmaca, Principal Investigator, Marmara University
Organization: Marmara University (Other)
Other Study IDs: MUPEDDENTNSL
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Malocclusion; Crossbite
Keywords: Removable Orthodontic Appliances; Clear Aligners; Oral Health-Related Quality of Life; Phonation; Anxiety; Visual Analog Scale (VAS)
MeSH Terms: conditions — Malocclusion; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with clear aligners: Patients aged between 6 and 12 years who required early orthodontic treatment and started clear aligner therapy were included in the study.
- Patients treated with removable orthodontic appliances: Patients aged between 6 and 12 years who required early orthodontic treatment and started removable orthodontic appliance therapy were included in the study.

SUMMARY:
This study aims to compare two different orthodontic treatment modalities-clear aligners and removable appliances-in children aged 6 to 12 years during the mixed dentition period. The primary focus of the research is to evaluate treatment-related changes in oral hygiene status, oral health-related quality of life, pain and anxiety levels, and speech function. By assessing multiple dimensions associated with early orthodontic intervention, the study seeks to provide a comprehensive understanding of how different appliance types influence clinical, functional, and psychosocial outcomes in pediatric patients.

DETAILED DESCRIPTION:
This study aims to compare two different orthodontic treatment modalities-clear aligners and removable appliances-in children aged 6 to 12 years during the mixed dentition period. The primary focus of the research is to evaluate treatment-related changes in oral hygiene status, oral health-related quality of life, pain and anxiety levels, and speech function. By assessing multiple dimensions associated with early orthodontic intervention, the study seeks to provide a comprehensive understanding of how different appliance types influence clinical, functional, and psychosocial outcomes in pediatric patients.

Detailed Description The mixed dentition period, occurring approximately between the ages of 6 and 12, represents a transitional developmental stage during which primary and permanent teeth coexist. In this phase, early diagnosis and treatment of orthodontic anomalies are particularly important to support functional, aesthetic, and psychosocial development and to minimize the need for more complex treatment in later stages.

Removable orthodontic appliances have traditionally been used to guide dental arch development, correct minor malocclusions, and eliminate harmful oral habits. Advances in digital technology have introduced clear aligners as an alternative treatment option that offers aesthetic and removable features. Despite their differences in design and material characteristics, both approaches are commonly used during early orthodontic treatment planning.

Orthodontic appliances may influence various aspects of oral function, including oral hygiene maintenance, periodontal health, caries risk, pain perception, anxiety levels, and speech performance. In growing children, treatment experiences may additionally shape cooperation, adaptation, and overall quality of life. Therefore, evaluating orthodontic interventions during the mixed dentition period requires consideration of not only mechanical efficiency but also broader functional and psychosocial parameters.

Appliance-related changes in intraoral volume and tongue movement can alter speech production, potentially affecting articulatory patterns and acoustic characteristics. Contemporary acoustic analysis methods, such as the use of specialized speech software, allow the objective measurement of frequency- and time-based acoustic parameters and provide complementary information to clinical observations.

This prospective study was designed to investigate how clear aligners and removable appliances influence oral hygiene status, pain and anxiety perception, oral health-related quality of life, and speech performance in children. Through standardized clinical assessments, validated questionnaires, and acoustic analysis, the study aims to generate multidimensional data that may guide clinical decision-making in early orthodontic treatment planning.

ELIGIBILITY:
Inclusion Criteria:

- Children aged between 6 and 12 years who applied to the Clinics of the Departments of Pedodontics and Orthodontics at Marmara University Faculty of Dentistry were included in the study.

* Patients were required to present with anterior cross-bite type malocclusion.
* Participants had to be cooperative, native Turkish speakers, and have no systemic disease, syndrome, craniofacial anomaly, or known allergy.
* Individuals with no apparent oro-facial anomaly, no hearing or speech impairment, and no reading or language difficulties were included.
* Based on clinical and radiographic evaluations, only patients whose malocclusions were determined to be dental in origin (not skeletal) were selected.
* Patients who did not require maxillary (palatal) expansion were also included in the study.

Exclusion Criteria:

* The study excluded patients who had severe periodontal disease, a history of systemic illness, a known allergy to any of the materials used in the study, poor oral hygiene, insufficient cooperation, or who did not agree to attend regular follow-up appointments during the study period.

Additionally, individuals with craniofacial anomalies or skeletal-origin malocclusions were not included. Participants with hearing impairments, non-native Turkish speakers, or those with any disease or history of surgery that could affect voice or speech quality were also excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consisted of systemically healthy children aged 6-12 years who presented to the Clinics of the Departments of Pediatric Dentistry and Orthodontics at Marmara University Faculty of Dentistry with an initial need for orthodontic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Formant frequencies (F1-F4) during speech production | At baseline (before treatment) and on the 1st, 3rd, 7th, and 14th days of treatment.
  Evaluation of phonation changes during early orthodontic treatment by analysing the first four formant frequencies (F1-F4) obtained from standardized speech recordings. Recordings were collected immediately before appliance placement and on days 1, 3, 7, and 14 after appliance insertion. Words selected from a standardized articulation test were read aloud by the participants, and acoustic data were analysed using Praat software to assess treatment-related variations in vowel resonance patterns.
  Units: Hertz (Hz)
  Higher values indicate:
  Changes in vowel resonance characteristics potentially related to treatment-related alterations in oral cavity configuration.

SECONDARY OUTCOMES:
Voice Onset Time (VOT) | At baseline (before treatment) and on the 1st, 3rd, 7th, and 14th days of treatment.
  Assessment of speech timing by measuring Voice Onset Time (VOT) from standardized speech recordings collected immediately before appliance placement and on days 1, 3, 7, and 14 after insertion. Selected words containing voiceless and voiced stop consonants were read aloud by participants, and VOT values were extracted using Praat software to evaluate treatment-related changes in articulatory timing.
  Units: Milliseconds (ms)
  Range:
  Approximately -100 ms to +150 ms (dependent on consonant type and participant characteristics)
  Higher values indicate:
  Longer delays between consonant release and onset of voicing, reflecting increased articulatory timing.
Spectral Centre of Gravity (CoG) | At baseline (before treatment) and on the 1st, 3rd, 7th, and 14th days of treatment.
  Assessment of spectral energy distribution during speech production by measuring the spectral Centre of Gravity (CoG) from standardized speech recordings. Recordings were obtained immediately before appliance placement and on days 1, 3, 7, and 14 after insertion. Selected words containing target consonants and vowels were read aloud by participants, and CoG values were extracted using Praat software to evaluate treatment-related changes in spectral balance and resonance characteristics.
  Units:Hertz (Hz) Range: Approximately 500-6000 Hz (dependent on sound type and participant characteristics) Higher values indicate: Spectral energy concentrated at higher frequencies, reflecting changes in resonance or articulatory configuration.
Spectral skewness | At baseline (before treatment) and on the 1st, 3rd, 7th, and 14th days of treatment.
  Assessment of spectral shape during speech production by measuring spectral skewness from standardized speech recordings. Recordings were obtained immediately before appliance placement and on days 1, 3, 7, and 14 after insertion. Selected words containing target consonants and vowels were read aloud by participants, and skewness values were extracted using Praat software to evaluate treatment-related changes in the asymmetry of the spectral energy distribution.
  Units: Dimensionless (no unit) Range: Approximately -3.0 to +3.0 (dependent on sound type and participant characteristics) Higher values indicate: Greater positive asymmetry of the spectral energy distribution (more energy concentrated above the mean frequency).
Spectral kurtosis | At baseline (before treatment) and on the 1st, 3rd, 7th, and 14th days of treatment.
  Assessment of spectral shape during speech production by measuring spectral kurtosis from standardized speech recordings. Recordings were obtained immediately before appliance placement and on days 1, 3, 7, and 14 after insertion. Selected words containing target consonants and vowels were read aloud by participants, and kurtosis values were extracted using Praat software to evaluate treatment-related changes in the peakedness of the spectral energy distribution.
  Units: Dimensionless (no unit) Range: Approximately -1.0 to +10.0 (dependent on sound type and participant characteristics) Higher values indicate: A more peaked spectral energy distribution with relatively more energy concentrated around the mean frequency.
Plaque Index (PI; Silness & Löe) | At baseline (before treatment) and 14th days of treatment.
  Assessment of dental plaque accumulation recorded at baseline, Day 1, and Day 14.
  Units: Score (0-3) Higher values indicate worse plaque accumulation.
Gingival Index (GI; Löe & Silness) | At baseline (before treatment) and 14th days of treatment.
  Evaluation of gingival inflammation recorded at baseline, Day 1, and Day 14. Units: Score (0-3) Higher values indicate worse gingival inflammation.
Pain perception (Visual Analog Scale) | 1st, 3rd, 7th, and 14th days of treatment
  Pain perception during early orthodontic treatment will be evaluated using a Visual Analog Scale (VAS). Participants will be asked to rate their pain on a 0-10 scale at multiple time points during adaptation to the appliance, including Days 1, 3, 7, and 14 following appliance insertion.
  Units: Scale score (0-10) Range: 0 (no pain) to 10 (severe pain)
  Higher values indicate:
  Greater perceived pain intensity.
Anxiety levels during treatment (State-Trait Anxiety Inventory for Children) | 1st, 3rd, 7th, and 14th days of treatment
  Anxiety levels during early orthodontic treatment will be evaluated using the State-Trait Anxiety Inventory for Children (STAI-C). Participants will complete the inventory on Days 1, 3, 7, and 14 following appliance insertion to assess treatment-related anxiety at multiple time points.
  Units: Scale score (20-60) Range: 20 (low anxiety) to 60 (high anxiety) Higher values indicate: Greater anxiety levels.
Oral health-related quality of life during treatment (OHIP-14) | 1st, 3rd, 7th, and 14th days of treatment
  Oral health-related quality of life during early orthodontic treatment will be evaluated using the Oral Health Impact Profile-14 (OHIP-14). Participants will complete the OHIP-14 questionnaire on Days 1, 3, 7, and 14 following appliance insertion to assess treatment-related changes in patient-reported oral health impact.
  Units: Scale score (0-56) Range: 0 (better oral health-related quality of life) to 56 (worse oral health-related quality of life) Higher values indicate: Worse oral health-related quality of life.

OTHER OUTCOMES:
Baseline oral health-related quality of life (COHIP-SF 19) | At baseline (before treatment)
  Baseline oral health-related quality of life will be assessed using the Child Oral Health Impact Profile Short Form (COHIP-SF 19) prior to appliance insertion.
  Units: Scale score (0-76) Range: 0 (better oral health-related quality of life) to 76 (worse oral health-related quality of life) Higher values indicate: Worse oral health-related quality of life.
Dental caries experience (DMFT/dft) | At baseline (before treatment)
  Baseline dental caries experience recorded prior to appliance insertion. Units: Number of teeth affected (0-28 depending on dentition) Higher values indicate more decayed, missing, and filled teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Atmaca, Doctor of Dental Surgery, Principal Investigator — Marmara Universty Faculty of Dentistry
Locations (1):
- Marmara Universty School of Dentistry, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including intraoral photographs and clinical evaluation scores) may be shared in scientific publications or presentations. Data will be limited to information relevant for scientific analysis and will not include any personal identifiers.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD), along with supporting documents such as the study protocol and statistical analysis plan, will be available beginning 6 months after publication of the primary study results and will remain available for 5 years following the publication date.
Access Criteria: Requests for access to de-identified individual participant data and supporting documents will be considered for academic or scientific research purposes. Interested researchers must submit a written proposal detailing the planned analysis, including objectives and statistical methods. Requests will be reviewed by the principal investigator and institutional review board (IRB) representatives to ensure ethical compliance and scientific merit. A data use agreement must be signed prior to data release. Requests can be submitted via email to the corresponding author listed in the publication.